CLINICAL TRIAL: NCT03269357
Title: Effectiveness of LARC Forward Contraceptive Counseling: LOWE - A Cluster Randomized Intervention Project
Brief Title: LARC Forward Counselling
Acronym: LOWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristina Gemzell Danielsson (Other)
Responsible Party: Sponsor-Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LoWe17
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Impact of Contraceptive Counselling on LARC Uptake and Unplanned Pregnancy
Keywords: LARC; contraception; counselling; unplanned pregnancy

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Clinics randomized to "intervention" will provide structured LARC centered counselling
  Interventions: Other: LARC forward structured contraceptive counselling
- Routine counselling (No Intervention): Clinics randomized to routine counselling

INTERVENTIONS:
Other: LARC forward structured contraceptive counselling — Training of health care providers (HCPs), use of information material and counselling tools
  Arms: Intervention

SUMMARY:
Training of health care providers and structured LARC forward counseling may contribute to increased LARC uptake. The hypothesis to be tested is that by introducing LARC forward counselling an increase in LARC usage will be the result as well as decreased unplanned pregnancy and abortion. It is expected that the results of this study will highlight the importance of LARC forward counseling and thus provide the evidence needed to train health care providers and increase access to LARC in youth clinics, midwifery clinics and for post abortion contraception.

ELIGIBILITY:
Inclusion Criteria:

* At risk for pregnancy (sexually active with men or anticipate becoming sexually active in the next 6 months).
* Do not desire pregnancy .
* No contraindications to LARC

Exclusion Criteria:

* Undergone tubal ligation or other sterilization procedure.
* Use of contraceptives for other purposes than contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
LARC prescriptions (recorded electronic prescriptions) | Evaluated at the index visit to the clinic
  The rate of women who receive a LARC prescription

SECONDARY OUTCOMES:
LARC placements recorded in patient records | Evaluated at 3months follow up (FU)
  The rate of women who has a LARC method placed following the baseline visit
Contraceptive method used reported by participants | Evaluated at 3,6 and 12 months FU
  The rate of women who use a contraceptive method
Satisfaction with the chosen contraceptive method reported by participants | Evaluated at 3,6 and 12 months FU
  Satisfaction with the prescribed contraceptive method
(Unplanned) pregnancy reported by participants and recorded in patient records | Evaluated at 3,6 and 12 months FU
  (Unplanned) pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- WHO centre, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwarsson KE, Podolskyi V, Bizjak I, Kallner HK, Gemzell-Danielsson K, Envall N. Effects of structured contraceptive counseling in young women: Secondary analyses of a cluster randomized controlled trial (the LOWE trial). Acta Obstet Gynecol Scand. 2024 Nov;103(11):2242-2251. doi: 10.1111/aogs.14954. Epub 2024 Sep 26. PMID 39327830
- [Derived] Emtell Iwarsson K, Larsson EC, Bizjak I, Envall N, Kopp Kallner H, Gemzell-Danielsson K. Long-acting reversible contraception and satisfaction with structured contraceptive counselling among non-migrant, foreign-born migrant and second-generation migrant women: evidence from a cluster randomised controlled trial (the LOWE trial) in Sweden. BMJ Sex Reprod Health. 2022 Apr;48(2):128-136. doi: 10.1136/bmjsrh-2021-201265. Epub 2022 Jan 31. PMID 35102001
- [Derived] Envall N, Emtell Iwarsson K, Bizjak I, Gemzell Danielsson K, Kopp Kallner H. Evaluation of satisfaction with a model of structured contraceptive counseling: Results from the LOWE trial. Acta Obstet Gynecol Scand. 2021 Nov;100(11):2044-2052. doi: 10.1111/aogs.14243. Epub 2021 Aug 25. PMID 34435347
- [Derived] Emtell Iwarsson K, Envall N, Bizjak I, Bring J, Kopp Kallner H, Gemzell-Danielsson K. Increasing uptake of long-acting reversible contraception with structured contraceptive counselling: cluster randomised controlled trial (the LOWE trial). BJOG. 2021 Aug;128(9):1546-1554. doi: 10.1111/1471-0528.16754. Epub 2021 Jun 7. PMID 33988917